CLINICAL TRIAL: NCT05659719
Title: A Pilot Project to Evaluate the Feasibility of Constructing a Concurrent External Control for Recifercept
Brief Title: A Study to Learn About Recifercept in Patients With Achondroplasia
Status: Completed | Type: Observational
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Other Study IDs: C4181010
Record Dates: First submitted 2022-10-12; First posted 2022-12-21 (Actual); Results first posted 2024-09-20 (Actual); Last update posted 2024-09-20 (Actual); Status verified 2024-05

CONDITIONS: Achondroplasia
MeSH Terms: conditions — Achondroplasia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective

GROUPS / COHORTS (2):
- Recifercept cohort: Achondroplasia patients enrolled in the recifercept phase 2 clinical trial
  Interventions: Other: Recifercept
- Natural history cohort: Achondroplasia patients enrolled in the achondroplasia natural history study

INTERVENTIONS:
Other: Recifercept — Patients received recifercept intervention in the phase 2 clinical trial
  Groups: Recifercept cohort

SUMMARY:
The purpose of this study is to learn about the study medicine (called recifercept) in people with achondroplasia. Achondroplasia is a very rare disease and patients of achondroplasia have short arms and legs. The study will include data already collected from a recifercept clinical trial and data collected from a separate study of achondroplasia. This study will compare patient experiences and will help the investigators determine if the study medicine, recifercept, is effective.

ELIGIBILITY:
Inclusion Criteria:

* All patients from Study C4181005 who have completed Visits 1 through 11 (at D183) will be included in this project.

To construct a concurrent external control, patients from Study C4181001 will need to meet the following inclusion criteria from Study C4181005 to be eligible for inclusion:

* Documented, confirmed genetic diagnosis of achondroplasia from historical medical records (test must have been performed at a laboratory fully accredited for genetic testing under local regulations)
* Aged ≥ 3 months to <11 years (up to the day before 11th birthday inclusive) at time of enrollment into the observational natural history study.
* Havecompleted at least 2 valid height/length measurements (at least 3 months apart)
* Assessed for Tanner stage 1 during physical examination before or at enrollment (must include assessment of breast development for females, testicular stage for males)
* Able to stand independently for height measurements (if ≥ 2 years of age at enrollment); If aged <2 years at enrollment, has a documented historical MRI brain/cervical spine performed in the previous 12 months.
* Have at least 6 months of available follow-up data after enrollment into the natural history study

Exclusion Criteria:

* Patients meeting any of the following criteria will not be included in the study:

  * Presence of severe obesity (BMI>95% percentile on Hoover-Fong BMI charts);
  * Body weight <7kg or >30kg
  * History of chronic kidney disease (CKD) or renal impairment
  * History of receipt of any treatment that are known to potentially affect growth (including oral steroids > 5 days in the last 6 months before enrollment, high dose inhaled corticosteroids (>800 mcg/day beclametasone equivalent) and medication for attention deficient hyperactivity disorder.
  * Less than 6 months since fracture or surgical procedure of any bone determined from the baseline visit date.
  * Presence of any internal guided growth plates/devices
  * History of removal of internal guided growth plates/devices within 6 months prior to enrollment

Ages: 3 Months to 10 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Achondroplasia patients, aged 3 months to 11 years old with documented and confirmed genetic diagnosis of achondroplasia, who have completed at least 2 valid height and length measurement in the natural history study and have at least 6 months of follow-up data in either the natural history study or the phase 2 recifercept trial.
Sampling Method: Probability Sample
Enrollment: 248 (Actual)
Dates: Start 2022-10-19 (Actual); Primary Completion 2023-05-16 (Actual); Study Completion 2023-05-16 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (1):
- Pfizer, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://pmiform.com/clinical-trial-info-request?StudyID=C4181010

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Data from eligible participants from C4181005 (NCT04638153) study and from C4181001 (NCT03794609) study were extracted and observed in this retrospective cohort study from 19-October-2022 to 16-May-2023 (approximately 7 months).
Groups:
- C4181005 Cohort: Recifercept 1 mg/kg QW: Eligible participants who received recifercept 1 milligram per kilogram (mg/kg) once weekly (QW) subcutaneously for 12 months in study C4181005 were included in this arm. Data from these participants were observed in this retrospective observational study.
- C4181005 Cohort: Recifercept 2 mg/kg BIW: Eligible participants who received recifercept 2 mg/kg twice weekly (BIW) subcutaneously for 12 months in study C4181005 were included in this arm. Data from these participants were observed in this retrospective observational study.
- C4181005 Cohort: Recifercept 1.5 mg/kg QD: Eligible participants who received recifercept 1.5 mg/kg once daily (QD) subcutaneously for 12 months in study C4181005 were included in this arm. Data from these participants were observed in this retrospective observational study.
- C4181001 Cohort: Eligible participants from study C4181001 who met the eligibility criteria for study C4181005 and had at least 6 months and up to 5 years follow-up data were included in this arm. Data from these participants were observed in this retrospective observational study.
Period: Overall Study
Arm/Group | C4181005 Cohort: Recifercept 1 mg/kg QW | C4181005 Cohort: Recifercept 2 mg/kg BIW | C4181005 Cohort: Recifercept 1.5 mg/kg QD | C4181001 Cohort
Started | 20 | 19 | 18 | 191
Completed | 20 | 19 | 18 | 2
Not Completed | 0 | 0 | 0 | 189
Not completed — At sponsor's request | 0 | 0 | 0 | 95
Not completed — Increased age moving to different baseline study with prospects of moving to intervention in future | 0 | 0 | 0 | 1
Not completed — Inclusion/Exclusion criteria | 0 | 0 | 0 | 5
Not completed — Wish of the child, or of the child's parent(S)/legal guardian(S), to withdrew from the study | 0 | 0 | 0 | 27
Not completed — Lost to Follow-up | 0 | 0 | 0 | 2
Not completed — Moved to another observational study | 0 | 0 | 0 | 1
Not completed — The child was enrolled in an interventional study | 0 | 0 | 0 | 55
Not completed — The child went to lower limbs elongation surgery in few weeks' time | 0 | 0 | 0 | 1
Not completed — The family wished to pursue a prescription a voxzogo instead of waiting for phase 3 | 0 | 0 | 0 | 2

BASELINE CHARACTERISTICS:
Population: Full Analysis set (FAS) included all enrolled participants who met the inclusion and exclusion criteria for the study and whose data was retrieved and observed in this study.
Groups:
- C4181005 Cohort: Recifercept 1 mg/kg QW: Eligible participants who received recifercept 1 mg/kg QW subcutaneously for 12 months in study C4181005 were included in this arm. Data from these participants were observed in this retrospective observational study.
- C4181005 Cohort: Recifercept 2 mg/kg BIW: Eligible participants who received recifercept 2 mg/kg BIW subcutaneously for 12 months in study C4181005 were included in this arm. Data from these participants were observed in this retrospective observational study.
- C4181005 Cohort: Recifercept 1.5 mg/kg QD: Eligible participants who received recifercept 1.5 mg/kg QD subcutaneously for 12 months in study C4181005 were included in this arm. Data from these participants were observed in this retrospective observational study.
- Total: Total of all reporting groups
Arm/Group | C4181005 Cohort: Recifercept 1 mg/kg QW | C4181005 Cohort: Recifercept 2 mg/kg BIW | C4181005 Cohort: Recifercept 1.5 mg/kg QD | C4181001 Cohort | Total
Number analyzed (Participants) | 20 | 19 | 18 | 191 | 248
Age, Continuous [Mean (Standard Deviation); unit: Years] | 5.75 (2.84) | 5.16 (2.59) | 5.83 (2.31) | 4.65 (2.59) | 4.86 (2.61)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9 | 9 | 6 | 79 | 103
  Male | 11 | 10 | 12 | 112 | 145
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3 | 0 | 2 | 10 | 15
  Not Hispanic or Latino | 16 | 19 | 15 | 181 | 231
  Unknown or Not Reported | 1 | 0 | 1 | 0 | 2
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race: White | 15 | 19 | 14 | 143 | 191
  Race: Black or African American | 0 | 0 | 0 | 2 | 2
  Race: Asian | 3 | 0 | 2 | 41 | 46
  Race: Other | 0 | 0 | 0 | 5 | 5
  Race: Multiracial | 1 | 0 | 1 | 0 | 2
  Race: Not reported | 1 | 0 | 1 | 0 | 2

OUTCOME MEASURES:

1. Primary Outcome: Mean Height Growth at Month 3
Description: Height growth was defined as ratio of observed change from baseline in standing height (centimeter) to expected change from baseline (centimeter) in reference population. For C4181001 cohort, baseline value was defined as the value recorded at the date of informed consent, whereas for C4181005 cohort the baseline value was the value taken at Day 1 before dosing.
Time Frame: Baseline, Month 3 [Eligible data extracted and observed in this retrospective cohort study from 19-October-2022 to 16-May-2023 (approximately 7 months)]
Population: FAS included all enrolled participants who met the inclusion and exclusion criteria for the study. Here, "Number of Participants Analyzed" signifies participants evaluable for this outcome measure.
Measure: Mean (Standard Deviation); unit: Ratio
Arm/Group | C4181005 Cohort: Recifercept 1 mg/kg QW | C4181005 Cohort: Recifercept 2 mg/kg BIW | C4181005 Cohort: Recifercept 1.5 mg/kg QD | C4181001 Cohort
Number analyzed (Participants) | 15 | 17 | 15 | 95
Ratio | 1.11 (0.487) | 0.84 (0.548) | 0.75 (0.707) | 1.07 (0.820)

2. Primary Outcome: Mean Height Growth at Month 6
Description: as for outcome 1
Time Frame: Baseline, Month 6 [Eligible data extracted and observed in this retrospective cohort study from 19-October-2022 to 16-May-2023 (approximately 7 months)]
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Ratio
Arm/Group | C4181005 Cohort: Recifercept 1 mg/kg QW | C4181005 Cohort: Recifercept 2 mg/kg BIW | C4181005 Cohort: Recifercept 1.5 mg/kg QD | C4181001 Cohort
Number analyzed (Participants) | 16 | 16 | 15 | 72
Ratio | 0.94 (0.429) | 1.06 (0.440) | 1.01 (0.453) | 1.11 (0.567)

3. Primary Outcome: Mean Height Growth at Month 9
Description: as for outcome 1
Time Frame: Baseline, Month 9 [Eligible data extracted and observed in this retrospective cohort study from 19-October-2022 to 16-May-2023 (approximately 7 months)]
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Ratio
Arm/Group | C4181005 Cohort: Recifercept 1 mg/kg QW | C4181005 Cohort: Recifercept 2 mg/kg BIW | C4181005 Cohort: Recifercept 1.5 mg/kg QD | C4181001 Cohort
Number analyzed (Participants) | 16 | 16 | 11 | 62
Ratio | 1.01 (0.374) | 0.97 (0.242) | 1.03 (0.285) | 1.10 (0.419)

4. Primary Outcome: Mean Height Growth at Month 12
Description: as for outcome 1
Time Frame: Baseline, Month 12 [Eligible data extracted and observed in this retrospective cohort study from 19-October-2022 to 16-May-2023 (approximately 7 months)]
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Ratio
Arm/Group | C4181005 Cohort: Recifercept 1 mg/kg QW | C4181005 Cohort: Recifercept 2 mg/kg BIW | C4181005 Cohort: Recifercept 1.5 mg/kg QD | C4181001 Cohort
Number analyzed (Participants) | 7 | 9 | 2 | 62
Ratio | 0.94 (0.298) | 1.06 (0.217) | 0.84 (0.036) | 1.10 (0.376)

5. Secondary Outcome: Mean Change From Baseline in Arm Span to Height/Length Difference at Months 3, 6, 9 and 12
Description: Arm span to standing height or length difference was defined as absolute value (arm length [centimeter] - standing height [centimeter]). For C4181001 cohort, baseline value was defined as the value recorded at the date of informed consent, whereas for C4181005 cohort the baseline value was the value taken at Day 1 before dosing.
Time Frame: Baseline, Months 3, 6, 9, 12 [Eligible data extracted and observed in this retrospective cohort study from 19-October-2022 to 16-May-2023 (approximately 7 months)]
Population: FAS included all enrolled participants who met the inclusion and exclusion criteria for the study. Here, "Number Analyzed" signifies participants evaluable for specific timepoints.
Measure: Mean (Standard Deviation); unit: Centimeter
Arm/Group | C4181005 Cohort: Recifercept 1 mg/kg QW | C4181005 Cohort: Recifercept 2 mg/kg BIW | C4181005 Cohort: Recifercept 1.5 mg/kg QD | C4181001 Cohort
Number analyzed (Participants) | 20 | 19 | 18 | 191
Centimeter
  Month 3: number analyzed (Participants) | 15 | 17 | 15 | 95
  Month 3 | 0.46 (0.956) | 0.02 (0.879) | -0.61 (1.705) | 0.09 (1.180)
  Month 6: number analyzed (Participants) | 16 | 16 | 15 | 72
  Month 6 | 0.19 (1.863) | 0.72 (1.028) | -0.47 (1.927) | 0.31 (1.706)
  Month 9: number analyzed (Participants) | 16 | 16 | 11 | 62
  Month 9 | 0.64 (0.890) | 0.69 (1.394) | 0.15 (0.781) | 0.53 (1.705)
  Month 12: number analyzed (Participants) | 7 | 9 | 2 | 61
  Month 12 | 0.47 (1.220) | 1.12 (1.754) | 0.20 (0.707) | 1.29 (3.745)

6. Secondary Outcome: Mean Change From Baseline in Knee Height: Lower Segment Ratio at Months 3, 6, 9 and 12
Description: Knee height: lower segment ratio was the ratio of knee to heel length to the difference between standing height and sitting height. For C4181001 cohort, baseline value was defined as the value recorded at the date of informed consent, whereas for C4181005 cohort the baseline value was the value taken at Day 1 before dosing.
Time Frame: as for outcome 5
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: Ratio
Arm/Group | C4181005 Cohort: Recifercept 1 mg/kg QW | C4181005 Cohort: Recifercept 2 mg/kg BIW | C4181005 Cohort: Recifercept 1.5 mg/kg QD | C4181001 Cohort
Number analyzed (Participants) | 20 | 19 | 18 | 191
Ratio
  Month 3: number analyzed (Participants) | 15 | 16 | 15 | 96
  Month 3 | -0.00 (0.020) | -0.01 (0.052) | 0.02 (0.037) | -0.09 (0.864)
  Month 6: number analyzed (Participants) | 16 | 15 | 14 | 72
  Month 6 | -0.00 (0.028) | -0.02 (0.062) | 0.00 (0.026) | -0.01 (0.048)
  Month 9: number analyzed (Participants) | 16 | 14 | 11 | 62
  Month 9 | -0.00 (0.027) | -0.02 (0.065) | 0.01 (0.026) | -0.01 (0.050)
  Month 12: number analyzed (Participants) | 7 | 8 | 2 | 62
  Month 12 | 0.00 (0.028) | -0.02 (0.081) | 0.02 (0.023) | -0.01 (0.049)

7. Secondary Outcome: Mean Change From Baseline in Height Standard Deviation Score (Z-Score) at Months 3, 6, 9, 12
Description: Z-score was calculated as the difference between mean observed standing height at specified visit and mean value of reference population divided by standard deviation of reference population. Z score indicated how similar the participant was to the reference population. A z-score of 0 is equal to the mean and is considered normal. Lower numbers indicate values lower than the mean and higher numbers indicate values higher than the mean. For C4181001 cohort, baseline value was defined as the value recorded at the date of informed consent, whereas for C4181005 cohort the baseline value was the value taken at Day 1 before dosing.
Time Frame: as for outcome 5
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: Z-score
Arm/Group | C4181005 Cohort: Recifercept 1 mg/kg QW | C4181005 Cohort: Recifercept 2 mg/kg BIW | C4181005 Cohort: Recifercept 1.5 mg/kg QD | C4181001 Cohort
Number analyzed (Participants) | 20 | 19 | 18 | 191
Z-score
  Month 3: number analyzed (Participants) | 15 | 17 | 15 | 96
  Month 3 | 0.03 (0.134) | -0.04 (0.173) | -0.02 (0.266) | 0.03 (0.289)
  Month 6: number analyzed (Participants) | 16 | 16 | 15 | 72
  Month 6 | -0.03 (0.205) | 0.03 (0.211) | -0.00 (0.236) | 0.06 (0.355)
  Month 9: number analyzed (Participants) | 16 | 16 | 11 | 62
  Month 9 | 0.00 (0.258) | -0.02 (0.214) | 0.02 (0.205) | 0.07 (0.412)
  Month 12: number analyzed (Participants) | 7 | 9 | 2 | 62
  Month 12 | -0.03 (0.327) | 0.07 (0.257) | -0.24 (0.169) | 0.12 (0.439)

8. Secondary Outcome: Number of Participants With Achondroplasia Related Orthopedic Complications
Description: Achondroplasia related orthopedic complications included lordosis, kyphosis, small foramen magnum: foramen magnum is slightly narrow and the spinal cord is slightly compressed at the level, foramen magnum stenosis, foramen magnum stenosis with associated c1-c2 secondary myelopathy, foramen magnum stenosis with mild posterior deformity of bulbospinal union, foramen magnum stenosis without spinal cord alteration, cervical myelomalacia; bulbar compression, marked stenosis of the foramen magnum with evident compression of bulb and bulb-medulla passage, mild foramen magnus stenosis, mild stenosis of foramen magnum, moderate to severe narrowing of the foramen magnum, severe stenosis at foramen magnum and stenosis foramen magnum.
Time Frame: C4181005 cohorts: 12 months; C4181001 cohort: 5 years [Eligible data extracted and observed in this retrospective cohort study from 19-October-2022 to 16-May-2023 (approximately 7 months)]
Population: FAS included all enrolled participants who met the inclusion and exclusion criteria for the study.
Measure: Count of Participants; unit: Participants
Arm/Group | C4181005 Cohort: Recifercept 1 mg/kg QW | C4181005 Cohort: Recifercept 2 mg/kg BIW | C4181005 Cohort: Recifercept 1.5 mg/kg QD | C4181001 Cohort
Number analyzed (Participants) | 20 | 19 | 18 | 191
Participants
  Lordosis | 0 | 0 | 0 | 79
  Kyphosis | 0 | 0 | 0 | 1
  Foramen magnum is slightly narrow | 0 | 0 | 0 | 1
  Foramen magnum stenosis | 0 | 0 | 0 | 3
  Foramen magnum stenosis with associated c1-c2 secondary myelopathy | 0 | 0 | 0 | 1
  Foramen magnum stenosis with mild posterior deformity of bulbospinal union | 0 | 0 | 0 | 1
  Foramen magnum stenosis without spinal cord alteration | 0 | 0 | 0 | 1
  Foramen magnum stenosis; cervical myelomalacia; bulbar compression | 0 | 0 | 0 | 1
  Marked stenosis of the foramen magnum with evident compression of Bulb and bulb-medulla passage | 0 | 0 | 0 | 1
  Mild foramen magnus stenosis | 0 | 0 | 0 | 1
  Moderate to severe narrowing of the foramen magnum | 0 | 0 | 0 | 1
  Severe stenosis at foramen magnum | 0 | 0 | 0 | 1
  Stenosis foramen magnum | 0 | 0 | 0 | 3

9. Secondary Outcome: Number of Participants With Other Achondroplasia Related Orthopedic Complications
Description: Other achondroplasia related orthopedic complications included otitis media, otitis media acute, hydrocephalus and obstructive sleep apnea syndrome.
Time Frame: as for outcome 8
Population: FAS included all enrolled participants who met the inclusion and exclusion criteria for the study.
Measure: Count of Participants; unit: Participants
Arm/Group | C4181005 Cohort: Recifercept 1 mg/kg QW | C4181005 Cohort: Recifercept 2 mg/kg BIW | C4181005 Cohort: Recifercept 1.5 mg/kg QD | C4181001 Cohort
Number analyzed (Participants) | 20 | 19 | 18 | 191
Participants
  Otitis media | 3 | 1 | 1 | 0
  Otitis media acute | 0 | 1 | 0 | 0
  Hydrocephalus | 0 | 0 | 0 | 2
  Obstructive sleep apnea syndrome | 0 | 1 | 0 | 0

ADVERSE EVENTS:
Time Frame: Not applicable as adverse events were not planned to be collected during this study.
Description: This observational retrospective study involved data that existed as structured data by the time of study start. In these data sources, individual participants data were not retrieved or validated. The minimum criteria for reporting an adverse event (AE) (i.e., identifiable participants, identifiable reporter, a suspect product, and event) was not met. Hence, AEs were not planned to be collected during the study and not reported.
Arm/Group | C4181005 Cohort: Recifercept 1 mg/kg QW | C4181005 Cohort: Recifercept 2 mg/kg BIW | C4181005 Cohort: Recifercept 1.5 mg/kg QD | C4181001 Cohort
All-Cause Mortality (participants affected / at risk) | 0/0 | 0/0 | 0/0 | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0 | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0 | 0/0 | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publication until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.

DOCUMENTS (2):
  • Study Protocol (2023-11-09): https://cdn.clinicaltrials.gov/large-docs/19/NCT05659719/Prot_000.pdf
  • Statistical Analysis Plan (2024-03-15): https://cdn.clinicaltrials.gov/large-docs/19/NCT05659719/SAP_001.pdf